CLINICAL TRIAL: NCT06292949
Title: Effect of Resistant Starch on Symptom Improvement and Intestinal Microbiome in Patients With Functional Constipation
Brief Title: Clinical Study of Resistant Starch in Improving Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huaping Xie (Other)
Responsible Party: Sponsor-Investigator, Huaping Xie, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TJ-IRB20230956
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Constipation
Keywords: Resistant starch; Gut microbiota
MeSH Terms: conditions — Constipation | interventions — Resistant Starch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistant starch intervention group (Experimental): or the recruited patients with functional constipation, stool samples were collected and 2 packets of resistant starch were taken every day, each packet of 10g. The resistant starch was brewed with 200ml warm water for 14 days, and the fecal samples of volunteers were collected on the 0th, 7th and 14th day. Patients filled out questionnaires on days 0 and 14 to evaluate the improvement of constipation symptoms.
  Interventions: Dietary Supplement: Resistant starch

INTERVENTIONS:
Dietary Supplement: Resistant starch — Constipated patients take 1 pack of resistant starch (20g/pack) daily for 14 days

SUMMARY:
Constipation is one of the most common gastrointestinal (GI) disorders in clinical practice, with approximately 11-20% of adults worldwide suffering from constipation. Clinically, the frequency of defecation is reduced, or the defecation is laborious, obstructed, difficult, and the stool is dry and difficult to solve, which is called constipation. Clinically, constipation is difficult to treat and over-reliance on laxatives often leads to water and electrolyte imbalance, gastrointestinal dysfunction, melanosis of the colon, relaxation of anal sphincter and other problems, and even leads to colorectal cancer, diabetes, anorexia nervosa and other complications in some cases. Therefore, it is very important to find a safe and effective laxative drug or diet to improve and relieve constipation symptoms. The health promotion effect of resistant starch is mainly due to the short-chain fat and gas produced by microbial fermentation in the colon, and its role in preventing colorectal cancer and some diet-related chronic diseases is stronger than dietary fiber, and it can effectively overcome the adverse odor, rough texture, poor quality and other drawbacks of food fortified with dietary fiber. Ruminococcus bromii is a specific microorganism that degrades resistant starch. The starch decomposing enzyme of R. bromii has a unique tissue structure and forms a multi-enzyme complex. Through the adhesion protein and dockerin module, it is attached to the cell surface through the scaffold protein in the cellulose body. Big data analysis showed that the relative abundance of R. bromii in healthy people was significantly higher than that in patients with constipation. Therefore, the purpose of this clinical trial is to supplement resistant starch to patients with constipation: (1) Observe whether the symptoms of patients with constipation have improved; (2) Analyze the changes of intestinal microorganisms in patients with constipation; and (3) Verify whether the relative abundance of R. bromii is increased and analyze the correlation between the relative abundance of R. bromii in intestine and the improvement of constipation symptoms in patients with constipation.

DETAILED DESCRIPTION:
Human intestinal microbiota is one of the densest microbial communities on earth, including highly diverse microbial communities, which provide metabolic, immune and protective functions and play a vital role in human health. Gastrointestinal microflora is affected by many factors, including genetics, host physiology (host age, disease, stress, etc.) and environmental factors, such as living conditions and drug use. At the same time, diet is considered to be a key environmental factor mediating gastrointestinal microflora composition and metabolic function . In view of the fact that it is difficult to be digested and absorbed by the human body, probiotics can enter the intestinal tract through the digestive tract, so as to improve intestinal microecology and promote lipid, protein and mineral metabolism.

Food rich in anti-digestible starch has many functions, such as controlling body weight, reducing blood lipids and blood sugar, regulating intestinal flora and so on, which has attracted the interest of many scholars and become a new field of international food research in recent years. Resistant starch (RS) is the anti-digestion part of compound polysaccharide starch. According to the conditions of enzymatic hydrolysis resistance and starch source, the digestible resistant starch was mainly divided into four types, namely RS1, RS2, RS3 and RS4. From the cause of resistance, RS1 and RS2 have natural resistance to amylase, and the resistance can disappear after gelatinization, while the resistance of RS3 and RS4 is formed by the transformation of starch in the process of food processing or food production. RS1 can coexist with RS2 or RS3 in the same kind of food, and the existence of RS4 can increase the food intake of RS3.

Only a small part of the digestible starch can be digested and absorbed in the small intestine, providing a very low utilization rate of glucose. When most of the rest of the undigested components enter the colon, they are fermented by the intestinal microflora, mainly producing short-chain fatty acids (SCFAs): acetate, propionate and butyrate. Although both acetate and propionate have health effects, butyrate is particularly thought to improve health and is the SCFA with the largest increase in RS intake. Butyrate plays an important role in human intestinal health, including reducing inflammation, reducing the risk of colon cancer and improving intestinal barrier function. In vivo and in vitro, resistant starch diet and butyrate significantly increased the proportion of ChAT immunoreactive intermuscular neurons, intestinal neurons expressed monocarboxylic acid transporter 2 (MCT2), small interference with RNA silenced MCT2, and prevented butyrate-induced increase in the proportion of ChAT immunoreactive neurons. Butyrate and trichostatin An increased the acetylation of histone H3 in intestinal neurons. Src signal pathway inhibitors can block the effect of butyrate. Resistant starch diet increased colonic transport, and butyrate increased cholinergic-mediated contraction of colonic circular muscles in vitro. Although RS has been shown to be one of the best fibers to increase butyrate levels in the population, it is clear that not everyone can get the same benefits, and some people do not respond to RS supplementation. This suggests that differences in individual microflora play an important role in determining the outcome of RS consumption, and we need to explore more deeply the mechanism of RS digestion and how it leads to the production of butyrate. In addition, more needs to be done to understand the health effects that may be affected by RS consumption beyond butyrate levels.

Due to the complex structure of RS, certain bacteria are required to initiate the degradation of this semi-crystalline material. R. bromii and Bifidobacterium juvenis are the only known human intestinal microorganisms with RS degrading ability.

R. bromii has received attention for its role as a keystone species for RS metabolism, feeding, and/or enabling other members of the gut microbiome to access this substrate. The starch-breaking enzyme of R. bromii has a unique organizational structure and forms a multi-enzyme complex, which is attached to the cell surface through the scaffold protein in the fibrinosomes through the adhesion protein and dockerin modules, so it is called amylasome. This system has been found in a variety of human rumenococcus, and the key enzyme structure of its amylasome is highly conserved across strains. Despite its incredible ability to degrade RS, R. bromii itself does not seem to outcompete or dominate other species, but rather serves a beneficial purpose by cross-feeding other species by releasing different lengths of sugars and acetate. One study found that median fecal butyrate increased by 50% after treatment with potato starch (RS2), but further examination of individual responses revealed different changes in butyrate. A follow-up study by the same group found that those with increased R. bromii abundance in their microbiota were more likely to have a higher butyrate response to potato starch, suggesting that the right combination of primary degrading bacteria and resistant starch is needed to increase butyrate production.

Constipation is one of the most common gastrointestinal (GI) disorders in clinical practice, with approximately 11-20% of adults worldwide suffering from constipation. Clinically, the frequency of defecation is reduced, or the defecation is laborious, obstructed, difficult, and the stool is dry and difficult to solve, which is called constipation [16]. Clinically, refractory constipation is difficult to treat and over-reliance on laxatives often leads to water and electrolyte imbalance, gastrointestinal dysfunction, melanosis of the colon, relaxation of anal sphincter and other problems, and even leads to colorectal cancer, diabetes, anorexia nervosa and other complications in some cases. Therefore, it is very important to find a safe and effective laxative drug or diet to improve and relieve constipation symptoms. The health promotion effect of resistant starch is mainly due to the short-chain fat and gas produced by microbial fermentation in the colon, and its role in preventing colorectal cancer and some diet-related chronic diseases is stronger than dietary fiber, and it can effectively overcome the adverse odor, rough texture, poor quality and other drawbacks of food fortified with dietary fiber. From the research data analysis point of view, as a natural, safe, "medicine and food" food resources, like dietary fiber, has a very important role in human health. It has important industrial application value and broad market development prospect, opens up a new field of functional food research, and makes up for the disadvantages of traditional dietary fiber.

In our previous analysis, stool microorganisms of 20 constipation patients and 20 healthy people were found to be very different in structure. The difference analysis indicated that Ruminococcus was abundant in healthy people. A classification model of AUROC0.967 was established using Lasso algorithm, and important features of the classification model were as follows: Ruminococcus is the feature with the highest weight. SPINGO notes that the genus Ruminococcus contains species, in which R. bromii has the highest relative abundance. A search of data from the GMrepo database revealed that Ruminococcus were found in 28,796 trials, belonging to 93 phenotypes. A total of 40,795 valid runs belonged to these phenotypes. The relative abundance of Ruminococcus in healthy people is significantly higher than that in constipated people, and the relative abundance of R. bromii in healthy people is significantly higher than that in constipated people. The relative abundance of Ruminococcus in healthy people was significantly higher than that in constipated people. Therefore, the purpose of this clinical trial is to supplement resistant starch for constipation patients and (1) observe whether the symptoms of constipation patients are improved; (2) To analyze the changes of intestinal microbes in patients with constipation; (3) Verify whether the relative abundance of R. bromii increases and analyze the correlation between the relative abundance of R. bromii in intestine and the improvement of constipation symptoms in patients with constipation.

The study was a non-randomized controlled study with no placebo group and enrolled 30 patients with functional constipation diagnosed by doctors. A questionnaire survey is used to understand whether the symptoms of constipation patients are improved. At the same time, stool samples are collected for metagenome sequencing analysis to study the changes of intestinal microbes of patients before and after the resistant starch intervention. Special attention is paid to whether the relative abundance of R. bromii is increased.

This study does not require recruitment advertisements, and subjects are recruited on a completely voluntary basis. Possible risks during the experiment are explained to subjects and informed consent is signed after they agree to join the study. The volunteers who agreed to join the experiment were surveyed by questionnaire to obtain their intestinal health and other health conditions, and screened according to the above research object selection criteria and exclusion criteria. The samples collected are named by the number, and the personal information of the subject will not be disclosed.The identity of the subjects was kept secret throughout the study, and only the number and disease phenotype were visible. Subjects may withdraw from the study at any time.

In this study, the composition and structure of the intestinal flora of the subjects will be analyzed, and the subjects can keep abreast of the progress of the test and analysis and obtain their own relevant data.

The resistant starch used in this study (HiMaize260) is produced by Ingredion. HI-MAIZE®260 resistant starch is a dietary fiber derived from Ingredion's proprietary high-amylose corn starch that enhances the nutritional content of everyday foods such as white bread, muffins, cookies, cakes and pasta.

The HI-MAIZE®260 standard is GB31637-2016, which conforms to the national standards for food safety. The HI-MAIZE®260 resistant starch contains approximately 53% resistant starch (dietary fiber) and 40% digestible starch and can be easily added to standard formulations by partially replacing plain flour. In addition, because HI-MAIZE®260 resistant starch contains fewer calories than flour, it enhances the nutritional content of food.

ELIGIBILITY:
Inclusion Criteria:

* The clinical manifestation is constipation, which meets the diagnostic criteria of Roman IV constipation.

Exclusion Criteria:

* Colonoscopy excludes patients with colorectal tumors within one or two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Changes in constipation symptoms | 14 days
  The results of the questionnaire filled out by the patients were collected and statistically analyzed, and the scores of constipation symptoms and PAC-QOL (patient assessment of constipation quality of life questionnaire) were tested by paired t-test. The higher the score, the more serious the constipation symptoms, and the lower the score means the relief of constipation symptoms. The minimum score of the scale is 0, the maximum score is 30, and a score of more than 15 can be regarded as constipation. The PAC-QOL is a specific scale for assessing the quality of life of patients with chronic constipation. The PAC-QOL consists of 28 items divided into four dimensions: worries and concerns (11 items), physical discomfort (4 items), psychological discomfort (8 items), and satisfaction (5 items). Each item was scored on a 5-point scale, and the more severe the illness, the higher the score.
Changes in the diversity of intestinal flora | 14 days
  To analyse changes in the diversity of intestinal flora before and after the administration of resistant starch in patients. Alpha diversity is a combination of species richness and evenness in a designated ecosystem. the Bray-Curtis distance reflects the variability in community composition and structure, with greater distances resulting in greater variability between communities.
Changes in the relative abundance of species of intestinal flora | 14 days
  To analyse the changes of relative abundance of species before and after the administration of resistant starch in patients.According to the species abundance table of each species, Krona analysis , relative abundance profile display, relative abundance cluster thermogram display, PCA and PCoA dimension reduction analysis, and Wilcoxon test of different species between groups were carried out.
Changes in the number of intestinal flora | 14 days
  Analyse the changes in the number of fecal flora before and after the administration of resistant starch in patients with constipation. In order to demonstrate more visually the changes in flora abundance after administration of resistant starch, statistical analyses were carried out using the number of patients who had a 1.5-fold increase or decrease in intestinal flora abundance before and after administration of resistant starch in all patients
Changes in the metabolic function of intestinal flora | 14 days
  According to the results of gene annotation, the ko gene family was mapped to KEGG database, and the annotation information of metabolic function was obtained, and the difference of metabolic function of fecal flora before and after taking resistant starch in constipation patients was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: ping h Xie, Study Chair — Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Department of Gastroenterology Tongji Hospital, Tongji Medical college, Huazhong University of Science and technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Questionnaires filled out by patients before and after taking resistant starch, and metagenomic sequencing results of stool samples

REFERENCES:
- [Result] Ni Y, Qian L, Siliceo SL, Long X, Nychas E, Liu Y, Ismaiah MJ, Leung H, Zhang L, Gao Q, Wu Q, Zhang Y, Jia X, Liu S, Yuan R, Zhou L, Wang X, Li Q, Zhao Y, El-Nezami H, Xu A, Xu G, Li H, Panagiotou G, Jia W. Resistant starch decreases intrahepatic triglycerides in patients with NAFLD via gut microbiome alterations. Cell Metab. 2023 Sep 5;35(9):1530-1547.e8. doi: 10.1016/j.cmet.2023.08.002. PMID 37673036
- [Result] Jumpertz R, Le DS, Turnbaugh PJ, Trinidad C, Bogardus C, Gordon JI, Krakoff J. Energy-balance studies reveal associations between gut microbes, caloric load, and nutrient absorption in humans. Am J Clin Nutr. 2011 Jul;94(1):58-65. doi: 10.3945/ajcn.110.010132. Epub 2011 May 4. PMID 21543530
- [Result] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Result] Goldsmith JR, Sartor RB. The role of diet on intestinal microbiota metabolism: downstream impacts on host immune function and health, and therapeutic implications. J Gastroenterol. 2014 May;49(5):785-98. doi: 10.1007/s00535-014-0953-z. Epub 2014 Mar 21. PMID 24652102
- [Result] Holscher HD. Dietary fiber and prebiotics and the gastrointestinal microbiota. Gut Microbes. 2017 Mar 4;8(2):172-184. doi: 10.1080/19490976.2017.1290756. Epub 2017 Feb 6. PMID 28165863
- [Result] Bach Knudsen KE, Laerke HN, Hedemann MS, Nielsen TS, Ingerslev AK, Gundelund Nielsen DS, Theil PK, Purup S, Hald S, Schioldan AG, Marco ML, Gregersen S, Hermansen K. Impact of Diet-Modulated Butyrate Production on Intestinal Barrier Function and Inflammation. Nutrients. 2018 Oct 13;10(10):1499. doi: 10.3390/nu10101499. PMID 30322146
- [Result] Zheng L, Kelly CJ, Battista KD, Schaefer R, Lanis JM, Alexeev EE, Wang RX, Onyiah JC, Kominsky DJ, Colgan SP. Microbial-Derived Butyrate Promotes Epithelial Barrier Function through IL-10 Receptor-Dependent Repression of Claudin-2. J Immunol. 2017 Oct 15;199(8):2976-2984. doi: 10.4049/jimmunol.1700105. Epub 2017 Sep 11. PMID 28893958
- [Result] Sindo T, Haga K, Yamamoto Y, Hayashi Y, Ozawa K. Studies on the interference between the allergic reactions caused by different antigen-antibody systems. Microbiol Immunol. 1978;22(8):509-13. doi: 10.1111/j.1348-0421.1978.tb00398.x. No abstract available. PMID 152836
- [Result] Venkataraman A, Sieber JR, Schmidt AW, Waldron C, Theis KR, Schmidt TM. Variable responses of human microbiomes to dietary supplementation with resistant starch. Microbiome. 2016 Jun 29;4(1):33. doi: 10.1186/s40168-016-0178-x. PMID 27357127
- [Result] Ze X, Duncan SH, Louis P, Flint HJ. Ruminococcus bromii is a keystone species for the degradation of resistant starch in the human colon. ISME J. 2012 Aug;6(8):1535-43. doi: 10.1038/ismej.2012.4. Epub 2012 Feb 16. PMID 22343308
- [Result] Ze X, Ben David Y, Laverde-Gomez JA, Dassa B, Sheridan PO, Duncan SH, Louis P, Henrissat B, Juge N, Koropatkin NM, Bayer EA, Flint HJ. Unique Organization of Extracellular Amylases into Amylosomes in the Resistant Starch-Utilizing Human Colonic Firmicutes Bacterium Ruminococcus bromii. mBio. 2015 Sep 29;6(5):e01058-15. doi: 10.1128/mBio.01058-15. PMID 26419877
- [Result] Mukhopadhya I, Morais S, Laverde-Gomez J, Sheridan PO, Walker AW, Kelly W, Klieve AV, Ouwerkerk D, Duncan SH, Louis P, Koropatkin N, Cockburn D, Kibler R, Cooper PJ, Sandoval C, Crost E, Juge N, Bayer EA, Flint HJ. Sporulation capability and amylosome conservation among diverse human colonic and rumen isolates of the keystone starch-degrader Ruminococcus bromii. Environ Microbiol. 2018 Jan;20(1):324-336. doi: 10.1111/1462-2920.14000. Epub 2017 Dec 7. PMID 29159997
- [Result] Crost EH, Le Gall G, Laverde-Gomez JA, Mukhopadhya I, Flint HJ, Juge N. Mechanistic Insights Into the Cross-Feeding of Ruminococcus gnavus and Ruminococcus bromii on Host and Dietary Carbohydrates. Front Microbiol. 2018 Nov 5;9:2558. doi: 10.3389/fmicb.2018.02558. eCollection 2018. PMID 30455672
- [Result] Cockburn DW, Koropatkin NM. Polysaccharide Degradation by the Intestinal Microbiota and Its Influence on Human Health and Disease. J Mol Biol. 2016 Aug 14;428(16):3230-3252. doi: 10.1016/j.jmb.2016.06.021. Epub 2016 Jul 6. PMID 27393306
- [Result] Baxter NT, Schmidt AW, Venkataraman A, Kim KS, Waldron C, Schmidt TM. Dynamics of Human Gut Microbiota and Short-Chain Fatty Acids in Response to Dietary Interventions with Three Fermentable Fibers. mBio. 2019 Jan 29;10(1):e02566-18. doi: 10.1128/mBio.02566-18. PMID 30696735
- [Result] Schiller LR. Chronic constipation: new insights, better outcomes? Lancet Gastroenterol Hepatol. 2019 Nov;4(11):873-882. doi: 10.1016/S2468-1253(19)30199-2. PMID 31609241
- [Result] Chang L, Di Lorenzo C, Farrugia G, Hamilton FA, Mawe GM, Pasricha PJ, Wiley JW. Functional Bowel Disorders: A Roadmap to Guide the Next Generation of Research. Gastroenterology. 2018 Feb;154(3):723-735. doi: 10.1053/j.gastro.2017.12.010. Epub 2017 Dec 27. PMID 29288656
- [Result] Annells M, Koch T. Older people seeking solutions to constipation: the laxative mire. J Clin Nurs. 2002 Sep;11(5):603-12. doi: 10.1046/j.1365-2702.2002.00626.x. PMID 12201887
- [Result] Cardin F, Minicuci N, Droghi AT, Inelmen EM, Sergi G, Terranova O. Constipation in the acutely hospitalized older patients. Arch Gerontol Geriatr. 2010 May-Jun;50(3):277-81. doi: 10.1016/j.archger.2009.04.007. Epub 2009 May 28. PMID 19481272
- [Result] Wallace C, Sinopoulou V, Gordon M, Akobeng AK, Llanos-Chea A, Hungria G, Febo-Rodriguez L, Fifi A, Fernandez Valdes L, Langshaw A, Saps M. Probiotics for treatment of chronic constipation in children. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD014257. doi: 10.1002/14651858.CD014257.pub2. PMID 35349168
- [Result] Koloski NA, Jones M, Wai R, Gill RS, Byles J, Talley NJ. Impact of persistent constipation on health-related quality of life and mortality in older community-dwelling women. Am J Gastroenterol. 2013 Jul;108(7):1152-8. doi: 10.1038/ajg.2013.137. Epub 2013 May 14. PMID 23670115
- [Result] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Result] Tian H, Ding C, Gong J, Ge X, McFarland LV, Gu L, Wei Y, Chen Q, Zhu W, Li J, Li N. Treatment of Slow Transit Constipation With Fecal Microbiota Transplantation: A Pilot Study. J Clin Gastroenterol. 2016 Nov/Dec;50(10):865-870. doi: 10.1097/MCG.0000000000000472. PMID 26751143

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT06292949/Prot_SAP_000.pdf